CLINICAL TRIAL: NCT06210958
Title: A Randomized Comparison of Cutaneous Sensory Blockade Between Ultrasound Guided Single and Triple Injections of Intertransverse Process Block in Patients Undergoing Video Assisted Thoracoscopic Surgery
Brief Title: Single- Vs. Triple-Injection Techniques for Intertransverse Process Blocks in Video-Assisted Thoracoscopic Surgery: a Randomized Trial on Sensory Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittitorn Supphapipat, Co-investigator, Department of Anesthesiology, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANE-2566-0137
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-01

CONDITIONS: Intertransverse Process Block; Video Assisted Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 2 groups: single injection of intertransverse process block and triple injection of intertransverse process block
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-group (Experimental): Single injection of ITPB at T4-5 level
  Interventions: Other: Intertransverse process block
- T-group (Experimental): Triple injection of ITPB at T3-4, T4-5, T5-6 levels
  Interventions: Other: Intertransverse process block

INTERVENTIONS:
Other: Intertransverse process block — The patients will be randomized into 2 groups which will receive the different techniques of the intertransverse process block

SUMMARY:
The intertransverse process block (ITPB) is an alternatives technique of regional anesthesia for thoracic surgery. However, the precise technique of ITPB remains developing. This study aims to evaluate the efficacy of ITPB injections which are single and triple injection in adult-patients undergoing video-assisted thoracoscopic surgery. The investigators hypothesize that cutaneous sensory block and perioperative pain outcomes including pain intensity and opioids consumption in patients who received triple injections of ITPB are better than that of single injection.

DETAILED DESCRIPTION:
Objectives: evaluate the efficacy of single and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for pulmonary resection Setting: Single center tertiary teaching hospital Participants: adult-patients who undergoing scheduled video-assisted thoracoscopic surgery for pulmonary resection.

Intervention: The patient will divide to 2 groups of intervention: single injection of ITPB (S-group) and triple injection of ITPB (T-group). The ITPB will be perform after routine general anesthesia. The primary outcomes is to compare the distribution of cutaneous block after single and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for pulmonary resection. The distribution of cutaneous block will be evaluate at PACU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20-70 years old
2. Undergoing scheduled the first time for each side of video-assisted thoracoscopic surgery (VATS) for pulmonary resection
3. American Society of Anesthesia (ASA) physical status I-III
4. Patients have ability to communicate and understand the study and accept to participate in study
5. Body weight >40 kg

Exclusion Criteria:

1. Patients who allergic to bupivacaine, lidocaine, NSAIDS, paracetamol, and dexamethasone
2. Patients who have following underlying disease: renal impairment (diagnosed of end-stage renal disease (ESRD) or chronic kidney disease (CKD) which estimated glomerular filtration rate (eGFR) < 60 ml/min per 1.73 square meters) , hepatic impairment (diagnosed of cirrhosis or evidence of abnormal liver function test which are increased liver enzymes or bilirubin level), coagulopathy (diagnosed of disease associated with abnormal coagulation, currently use any anticoagulants or evidence of prolong prothrombin time (PT) or partial thromboplastin time (PTT)), thrombocytopenia (platelet count less than 150,000/microliter), platelet disfunction from any causes such as current use antiplatelet or uremia (BUN level > 60 mg/dL) , morbid obesity (BMI >40 kg/m2), pre-existing neurological deficits, chronic pain (diagnosed of chronic pain disease or current use regular analgesic drugs), or any drug addiction • Withdrawal criteria: a participant will be withdrawn from the study in case of

1. Procedural failure: the operator cannot place the needle tip in the intertransverse tissue according to the technical difficulty or abnormal anatomy after 15 minutes of performing the block (from the beginning of needle insertion to the injection of local anesthetic) 2. Anesthetic related events including cardiac arrest, difficult intubation 3. Surgical related events including massive bleeding, major organ injury, converted operation to open thoracotomy and reoperation within admission 4. Participant related reasons including patient's willing to withdraw from the study or failure to adhere adequately to protocol requirements such as premature discharge. However, the withdrawn participant will be continued follow up of clinical outcome.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To compare the distribution of cutaneous block after the inter transverse process block and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for lobectomy | at 1 hour after the end of surgery
  the distribution of cutaneous block is the cutaneous sensory distribution of dermatomes involvement by the intertransverse process block. A cutaneous sensory distribution is defined as an area of reduced sensitivity to cold touch as compare to the abdomen which participants know as 'normal'. The assessment begins at the mid-clavicular line on the block side, processing laterally to the posterior axillary line on the chest wall and apex of axilla (between T2-T10 dermatomes) at about 1-cm intervals, bilaterally.

SECONDARY OUTCOMES:
To compare pain intensity using numerical rating scale during the first 24-hours postoperative period after single and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for lobectomy | 24 hour after surgery
  The numerical rating scale is a pain scales using numbers from 0 to 10. A score of 0 means no pain, and 10 means the worst pain.
To compare opioids consumption during the intraoperative and the first 24-hours postoperative period after single and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for lobectomy | 24 hour after surgery
To compare adverse complication (pneumothorax, hemothorax) after single and triple injections of ultrasound-guided ITPB in adult patients undergoing video-assisted thoracoscopic surgery for lobectomy | 24 hour after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kittitorn Supphapipat, Principal Investigator — Department of Anesthesiology, Faculty of Medicaine, Chaing Mai University
Locations (1):
- Department of Anesthesiology, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared

REFERENCES:
- [Background] Bade BC, Dela Cruz CS. Lung Cancer 2020: Epidemiology, Etiology, and Prevention. Clin Chest Med. 2020 Mar;41(1):1-24. doi: 10.1016/j.ccm.2019.10.001. PMID 32008623
- [Background] Sihoe ADL. Video-assisted thoracoscopic surgery as the gold standard for lung cancer surgery. Respirology. 2020 Nov;25 Suppl 2:49-60. doi: 10.1111/resp.13920. Epub 2020 Jul 30. PMID 32734596
- [Background] Jones GS, Baldwin DR. Recent advances in the management of lung cancer. Clin Med (Lond). 2018 Apr 1;18(Suppl 2):s41-s46. doi: 10.7861/clinmedicine.18-2-s41. PMID 29700092
- [Background] Marshall K, McLaughlin K. Pain Management in Thoracic Surgery. Thorac Surg Clin. 2020 Aug;30(3):339-346. doi: 10.1016/j.thorsurg.2020.03.001. Epub 2020 Apr 29. PMID 32593366
- [Background] Tong Y, Wei P, Wang S, Sun Q, Cui Y, Ning N, Chen S, He X. Characteristics of Postoperative Pain After VATS and Pain-Related Factors: The Experience in National Cancer Center of China. J Pain Res. 2020 Jul 21;13:1861-1867. doi: 10.2147/JPR.S249134. eCollection 2020. PMID 32765060
- [Background] Takenaka S, Saeki A, Sukenaga N, Ueki R, Kariya N, Tatara T, Hirose M. Acute and chronic neuropathic pain profiles after video-assisted thoracic surgery: A prospective study. Medicine (Baltimore). 2020 Mar;99(13):e19629. doi: 10.1097/MD.0000000000019629. PMID 32221089
- [Background] Zhang Y, Zhou R, Hou B, Tang S, Hao J, Gu X, Ma Z, Zhang J. Incidence and risk factors for chronic postsurgical pain following video-assisted thoracoscopic surgery: a retrospective study. BMC Surg. 2022 Mar 2;22(1):76. doi: 10.1186/s12893-022-01522-1. PMID 35236334
- [Background] Peng J, Wang Z, Ma L, Ma W, Liu G, Zhang H, Wang Q, Zhu B, Zhao L. Incidence and Influencing Factors of Chronic Postthoracotomy Pain in Lung Tumor Patients. J Healthc Eng. 2022 Feb 24;2022:7584481. doi: 10.1155/2022/7584481. eCollection 2022. PMID 35251576
- [Background] Piccioni F, Ragazzi R. Anesthesia and analgesia: how does the role of anesthetists changes in the ERAS program for VATS lobectomy. J Vis Surg. 2018 Jan 11;4:9. doi: 10.21037/jovs.2017.12.11. eCollection 2018. PMID 29445595
- [Background] Bugada D, Lorini LF, Lavand'homme P. Opioid free anesthesia: evidence for short and long-term outcome. Minerva Anestesiol. 2021 Feb;87(2):230-237. doi: 10.23736/S0375-9393.20.14515-2. Epub 2020 Aug 4. PMID 32755088
- [Background] Nafziger AN, Barkin RL. Opioid Therapy in Acute and Chronic Pain. J Clin Pharmacol. 2018 Sep;58(9):1111-1122. doi: 10.1002/jcph.1276. Epub 2018 Jul 9. PMID 29985526
- [Background] Olausson A, Svensson CJ, Andrell P, Jildenstal P, Thorn SE, Wolf A. Total opioid-free general anaesthesia can improve postoperative outcomes after surgery, without evidence of adverse effects on patient safety and pain management: A systematic review and meta-analysis. Acta Anaesthesiol Scand. 2022 Feb;66(2):170-185. doi: 10.1111/aas.13994. Epub 2021 Nov 11. PMID 34724195
- [Background] Feray S, Lubach J, Joshi GP, Bonnet F, Van de Velde M; PROSPECT Working Group *of the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guidelines for video-assisted thoracoscopic surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2022 Mar;77(3):311-325. doi: 10.1111/anae.15609. Epub 2021 Nov 5. PMID 34739134
- [Background] Lin J, Liao Y, Gong C, Yu L, Gao F, Yu J, Chen J, Chen X, Zheng T, Zheng X. Regional Analgesia in Video-Assisted Thoracic Surgery: A Bayesian Network Meta-Analysis. Front Med (Lausanne). 2022 Apr 6;9:842332. doi: 10.3389/fmed.2022.842332. eCollection 2022. PMID 35463038
- [Background] Richardson J, Lonnqvist PA. Thoracic paravertebral block. Br J Anaesth. 1998 Aug;81(2):230-8. doi: 10.1093/bja/81.2.230. No abstract available. PMID 9813528
- [Background] Sharma R, Louie A, Thai CP, Dizdarevic A. Chest Wall Nerve Blocks for Cardiothoracic, Breast Surgery, and Rib-Related Pain. Curr Pain Headache Rep. 2022 Jan;26(1):43-56. doi: 10.1007/s11916-022-01001-5. Epub 2022 Jan 28. PMID 35089532
- [Background] Kim SH. Anatomical classification and clinical application of thoracic paraspinal blocks. Korean J Anesthesiol. 2022 Aug;75(4):295-306. doi: 10.4097/kja.22138. Epub 2022 Apr 4. PMID 35368174
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Junior Ade P, Erdmann TR, Santos TV, Brunharo GM, Filho CT, Losso MJ, Filho GR. Comparison between continuous thoracic epidural and paravertebral blocks for postoperative analgesia in patients undergoing thoracotomy: Systematic review. Braz J Anesthesiol. 2013 Sep-Oct;63(5):433-42. doi: 10.1016/j.bjane.2013.10.002. Epub 2013 Nov 19. PMID 24565302
- [Background] Cho TH, Kwon HJ, O J, Cho J, Kim SH, Yang HM. The pathway of injectate spread during thoracic intertransverse process (ITP) block: Micro-computed tomography findings and anatomical evaluations. J Clin Anesth. 2022 May;77:110646. doi: 10.1016/j.jclinane.2022.110646. Epub 2022 Jan 10. PMID 35021139